CLINICAL TRIAL: NCT07187271
Title: Comparison of Respiratory Parameters, Aerobic Capacity, and Sleep Quality in Individuals With Thoracic Adolescent Idiopathic Scoliosis
Brief Title: Assessment of Respiratory Parameters, Aerobic Capacity and Sleep Quality in Thoracic AIS
Status: Not yet recruiting | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Gizem Sevindi, Physiotherapist, Uskudar University
Other Study IDs: 2025-PT-GIZEM-AIS; 61351342/020-774 (Other: USKUDAR UNIVERSITESI GIRISIMSEL OLMAYAN ARASTRIMALAR ETIK KURULU BASKANLIGI); 2025-05/36 (Other: ACIBADEM MEHMET ALI AYDINLAR UNIVERSIRTESI TIBBI ARASTIRMALAR DEGERLENDIRME KURULU)
Record Dates: First submitted 2025-09-19; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: AIS; ISST classification; Thoracic AIS; Thoracolumbar AIS; Cobb angle; Angle of Trunk Rotation (ATR); Pulmonary function test; FEV1; FVC; Respiratory muscle strength; MIP (Maximal Inspiratory Pressure); MEP (Maximal Expiratory Pressure); Aerobic capacity; Incremental Shuttle Walk Test (ISWT); PUKİ (Pittsburgh Sleep Quality Index); SAQ (Scoliosis Appearance Questionnaire)
MeSH Terms: conditions — Laurin-Sandrow syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T-Type: Participants diagnosed with thoracic type Adolescent Idiopathic Scoliosis (AIS), defined as a primary thoracic curve according to ISST classification. Eligible individuals are between 12 and 20 years of age and meet the inclusion criteria. All outcome measures, including pulmonary function tests, respiratory muscle strength, aerobic capacity, sleep quality, and body image assessments, will be evaluated in this group.
- TL-Type: Participants diagnosed with thoracolumbar type Adolescent Idiopathic Scoliosis (AIS), defined as a primary thoracolumbar curve according to ISST classification. Eligible individuals are between 12 and 20 years of age and meet the inclusion criteria. All outcome measures, including pulmonary function tests, respiratory muscle strength, aerobic capacity, sleep quality, and body image assessments, will be evaluated in this group.

SUMMARY:
This study aims to compare respiratory parameters -including pulmonary function and respiratory muscle strength-as well as aerobic capacity and sleep quality in individuals with thoracic adolescent idiopathic scoliosis. Participants will be categorized according to the ISST classification into T-type and TL-type curvature patterns. The study will evaluate differences between these groups using standardized clinical assessments.

DETAILED DESCRIPTION:
This study aims to compare respiratory parameters (including pulmonary function tests and respiratory muscle strength), aerobic capacity, and sleep quality in individuals aged 12 to 20 years with thoracic adolescent idiopathic scoliosis (AIS), classified as T-type or TL-type based on the ISST classification. The study will be conducted at the Spine Health Center of Acıbadem Maslak Hospital.

A total of 30 volunteer participants will be included. Sagittal plane curvatures will be assessed using EOS imaging, and Cobb angles and axial trunk rotation (ATR) will be recorded. ATR will be measured using a scoliometer during the Adams forward bend test. Demographic data including age, sex, height, weight, and dominant side will also be collected.

Pulmonary function will be assessed using FVC and FEV₁ measurements, while respiratory muscle strength will be evaluated using the Cosmed Pony Fx device to measure maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP). Each test will be repeated three times, and the highest value will be used for analysis. Aerobic capacity will be evaluated using a progressive shuttle walk test. Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), and body image perception will be evaluated using the Scoliosis Appearance Questionnaire.

This is a cross-sectional observational study. Data will be compared between the T-type and TL-type scoliosis groups. The study will be supported by Üsküdar University, and all required devices will be provided by the university.

ELIGIBILITY:
Inclusion Criteria:

Individuals with a Cobb angle greater than 10 degrees Adolescents aged 12-20 years diagnosed with thoracic Adolescent Idiopathic Scoliosis, classified as T-type or TL-type according to ISST classification Patients currently undergoing brace treatment

Exclusion Criteria:

Individuals with a history of spinal surgery Individuals with neurological disorders Individuals with a diagnosed psychiatric disorder Pregnant individuals Individuals who do not provide consent to participate in the study

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent patients aged 12-20 years with thoracic or thoracolumbar Adolescent Idiopathic Scoliosis recruited from Acıbadem Maslak Hospital Spine Health Center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-05 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Strength (MIP, MEP) | At baseline (single measurement during study enrollment)
  Respiratory muscle strength will be assessed using an electronic mouth pressure meter (Cosmed Pony FX, ) by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP). This outcome evaluates the strength of inspiratory and expiratory muscles in participants with thoracic and thoracolumbar AIS.

SECONDARY OUTCOMES:
Pulmonary Function (FVC, FEV₁) | At baseline (single measurement during study enrollment)
  Pulmonary function will be assessed using an electronic spirometry device (Cosmed Pony FX, ) by measuring Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 second (FEV₁). This outcome evaluates respiratory capacity in participants with thoracic and thoracolumbar AIS.
Aerobic Capacity (Incremental Shuttle Walk Test, ISWT) | At baseline (single measurement during study enrollment)
  Aerobic capacity will be measured using the Incremental Shuttle Walk Test (ISWT) to determine exercise tolerance and endurance in participants with thoracic and thoracolumbar AIS.
Sleep Quality (PUKI - Pittsburgh Sleep Quality Index) | At baseline (single measurement during study enrollment)
  Sleep quality will be evaluated with the validated Turkish version of the Pittsburgh Sleep Quality Index (PUKI). Higher scores indicate poorer sleep quality.
Body Image (Scoliosis Appearance Questionnaire, SAQ) | At baseline (self-administered questionnaire during study enrollment)
  Body image perception will be assessed with the Scoliosis Appearance Questionnaire (SAQ) to evaluate patients' perception of spinal deformity.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Eyüboğlu, PhD., Study Director — Uskudar University; Mert İlhan, MSc., Principal Investigator — Uskudar University; Gizem Sevindi, PT., Principal Investigator — Uskudar University; Çağlar Yılgör, Prof., Principal Investigator — Koç University
Locations (1):
- Acıbadem Hospital, Istanbul, Europe & Central Asia - Upper Middle Income, Turkey (Türkiye)